CLINICAL TRIAL: NCT04791618
Title: Impact of Technology-based Intervention for Improving Self-management Behaviors in Black Adults; Sub-project of Biological and Socio-cultural Determinants and Management of Cardiovascular Health Factors in Multi-ethnic Populations
Brief Title: MECA Clinical Intervention ( MECA Health360x)
Acronym: MECAH360x
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Morehouse School of Medicine (Other)
Collaborators: Emory University (Other)
Responsible Party: Principal Investigator, Priscilla Pemu, Professor, Morehouse School of Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 809392
Record Dates: First submitted 2017-10-09; First posted 2021-03-10 (Actual); Last update posted 2021-03-10 (Actual); Status verified 2021-03

CONDITIONS: Cardiovascular Health; Self-management
Keywords: Cardiovascular health risk; e-health lifestyle intervention; ehealthystrides; Life simple 7; Health coach; Health equity; Behavioral intervention; Hypertension; Obesity; Diabetes Mellitus; Helath360x; Tobacco use
MeSH Terms: conditions — Hypertension; Obesity; Diabetes Mellitus; Tobacco Use | interventions — Organizational Objectives

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Health360x only (High tech) (Active Comparator): Access to Health360x technology only for 6 months Behavioral: Health360x Participants will receive Access to health360x which provides monitoring, in the moment color coded feedback and goal setting for self- management skills. Every participant will view an orientation video which will include information on how to access Health360 from home and other internet connected devices; how to use activity monitors provided by the study and sphygmomanometer. They will receive an introduction to heart health curriculum, quizzes and discussion forums. Participants will be encouraged to upload their data at least once a week and to access the curriculum as often as desired. Technological and customer service support related to use of the Helath360x application will be available online and by phone.
  The Health360x application will send messages to participants in this arm reminding them to perform study related activities.
  Interventions: Behavioral: Health360x only (High tech)
- Health360x plus Coach (High tech High touch) (Experimental): Health360x technology plus health coach Behavioral: Health360x plus health coach Participants will receive all of the resources in Arm A and Health coach interactions.
  The Health coach will send messages to participants in this arm reminding them to perform study related activities. The coach interactions will be focused on helping with attainment of self- management behaviors
  Interventions: Behavioral: Health360x plus health coach; Behavioral: Health360x only (High tech)

INTERVENTIONS:
Behavioral: Health360x plus health coach — Access to health360x which provides monitoring, in the moment color coded feedback and goal setting for self management skills
  Other Names: Health coach intervention; Self management skills training; Goal setting; Monitoring; Healthy coping
  Arms: Health360x plus Coach (High tech High touch)
Behavioral: Health360x only (High tech) — All participants will have access to Helath360x with reminders generated for goal setting.
  Other Names: e-Health lifestyle intervention; Self management skills training; Goal setting; Monitoring; Healthy coping

SUMMARY:
The purpose of this research is to test whether a technology application(Health360x) that lets participants set goals for better health and track health can help participants reduce their heart disease risk. Investigators will compare life style intervention using Health360x alone with Health360xs plus health coach on AHA(American Heart Association) LS7 scores after 6 months.

DETAILED DESCRIPTION:
Study volunteers' participation in this study will last for 6 months. Investigators will ask participants to examine their own health behaviors. The purpose of the examination is to find the areas that need improvement so participants can work on them. Investigators will use technology in the form of Health360x to support participant efforts to change health behaviors.

This list below, shows the activities you will perform as part of this research.

Arm A ='High tech' Arm B='High tech high touch"

1. Recruitment Phone call: During this call, investigators will do the following:

   * Collect email address
   * Phone# that can receive text messages
   * Contact information for 2 close friends/relatives
2. Investigators will email participants enrollment and welcome package that contains links to the

   * Online screening form
   * Consent form Please complete both forms
3. Investigators will send participants a link to online training videos and Health360x user manual that show how to use health360x and the online user manual

   • Participants will show investigative team that they know how to use Health360x by completing a proficiency test
4. Investigators will have Live chat sessions to answer questions about the project by the health coach and PI. Participants can access these as needed
5. Participants will be assigned by chance, to High tech only(Arm A) or high tech and high touch(Arm B). Participant will receive an email notification of what study arm they are enrolled in
6. Self- assessment; LS7 score
7. Participant will receive a sleep/activity tracker; Investigators will work to obtain a Blood Pressure monitor through participants' usual health insurance
8. Weekly goal setting; personal action plan x4 weeks Arm A participants will receive email prompts to complete. Arm B participants will complete; 45minute-1 hour meetings with health coach (recorded)
9. Every 2-week goal setting; personal action plans x4 Arm A participants will receive email prompts to complete; Arm B participants will complete 45 minute-1 hour long meetings with health coach(recorded)
10. Every 1 monthly goal setting; personal action plan x3 Arm A participants will receive email prompts to complete; Arm B participants will complete 45 minute-1 hour long meetings with health coach(recorded)

ELIGIBILITY:
Inclusion Criteria:

* Already participating in baseline clinical study
* Volunteers with AHA LS7 scores of 4 or lower who have access to internet (community or personal),self-reported ability to participate in physical activity, and English fluency.

Exclusion Criteria:

* CAD documented by CAD diagnosis or prior acute myocardial infarction, percutaneous coronary intervention, coronary artery bypass surgery, or chronic angina; aortic stenosis; inability to participate in increased physical activity; history of alcohol or drug abuse or psychiatric diagnosis that would interfere with ability to participate.

Pregnant and/or breastfeeding women will be excluded. Cognitive deficits severe enough to preclude participation or any medical or surgical problem that precludes meaningful participation; unwillingness to use the internet

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2017-05-01 (Actual); Primary Completion 2020-09-30 (Actual); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Life Simple 7(LS7 the metrics for defining ideal cardiovascular health) score at 6-month follow-up | 6 months
  The LS7 score consists of 4 behavioral and 3 clinical measures. The behavioral measures are smoking, body Mass Index (BMI), physical activity and healthy dietary pattern. The clinical measures are blood pressure, total cholesterol and fasting plasma glucose.Each LS7 component will be given a point score of 0, 1, or 2 to represent poor, intermediate, or ideal health, respectively. Then, an overall LS7 score ranging from 0 to 14 will be calculated as the sum of the LS7 component scores. The overall LS7 score will be further classified as inadequate (0-4), average (5-9), or optimum (10-14) cardiovascular health.

SECONDARY OUTCOMES:
Self management skills acquired | 6 months
  Self management skills are patterned on the AADE 7 self care behaviors. A skill is acquired when the participant reports a score of 7 or higher on a 10-point scale.
  Healthy Coping Healthy Eating Being Active Monitoring Taking Medication Problem Solving Reducing Risks
Change in Systolic Blood Pressure: | Baseline, Month 6
  Blood pressure readings will be made three times with the subject at rest in the sitting position using a cuff of the appropriate size and a standardized procedure. The average of the three systolic blood pressure measurements will be calculated. Blood pressure will be categorized according to Joint National Committee recommendations.
Change in Diastolic Blood Pressure | Baseline, Month 6
  Blood pressure readings will be made three times with the subject at rest in the sitting position using a cuff of the appropriate size and a standardized procedure. The average of the three diastolic blood pressure measurements will be calculated. Blood pressure will be categorized according to Joint National Committee recommendations.
Change in Delta Nutrition Intervention Research Initiative Food Frequency Questionnaire (Delta NIRI FFQ) | Baseline, Month 6
  Dietary intake of fruits and vegetables will be assessed using the Lower Mississippi Delta Nutrition Intervention Research Initiative food frequency questionnaire (Delta NIRI FFQ). The Delta NIRI FFQ is a 283-item, interviewer administered questionnaire that asks if respondents have had certain food items in the past 24 hours, including foods that are commonly consumed in the southern United States.
Change in Blood Glucose | Baseline, Month 3, Month 6
  Blood glucose will be measured as milligrams per deciliter at Baseline, 3 months after the start of the intervention and at the end of the intervention at month 6. Normal, fasting blood glucose levels are between 70 to 100 mg/dL.
Change in Distance Walked Daily | Baseline, Month 3, Month 6
  The total distance walked daily in miles will be measured by a pedometer or the exercise application for mobile devices.
Change in Short Form-12 Health Survey Questionnaire (SF-12) score | Baseline, Month 3, Month 6
  The Short Form-12 Health Survey Questionnaire (SF-12) is a measure of general physical and mental health.
  The SF-12 consists of 12 items with a Likert-type response format that measures quality of life with a Physical Component Summary (PCS) and Mental Component Summary (MCS). Subscales associated with the PCS include physical functioning, role limitations due to physical problems, bodily pain, and general health perceptions. Subscales associated with the MCS include vitality (energy and fatigue), social functioning, role limitations due to emotional problems, and mental health. The total score for each subscale ranges from 0 to 100 and low values represent a poor health state while high values represent a good health state.
Change in Stress Management | Baseline, then monthly through Month 6
  Participants will report on their stress management monthly via free text responses in an online format.
Change in Weight | Baseline, then monthly through Month 6
  Participants will report their weight in pounds once per month during the intervention period.
Change in Tobacco Use | Baseline, then monthly through Month 6
  Participants will report whether or not they have used tobacco once per month during the intervention period.

OTHER OUTCOMES:
Change in High-sensitivity C-reactive Protein (HsCRP) | Baseline, Month 6
  C-reactive protein (CRP) is a biomarker of cardiovascular health which increases in the blood when inflammation is present. The Hs-CRP test can measure low levels of CRP which indicate the risk of developing cardiovascular disease (CVD). A measurement of less than 1.0 milligrams of CRP per liter of blood (mg/L) is defined as low risk, 1.0 to 3.0 mg/ L is average risk, and above 3.0 mg/L is high risk of developing CVD
Change in Plasma Cysteine | Baseline, Month 6
  Plasma cysteine is a biomarker of oxidative stress, which is implicated in the pathophysiology of multiple conditions including cardiovascular disease (CVD). Higher levels of cysteine are associated with increased risk of CVD.
Change in Cystine | Baseline, Month 6
  Cystine is the oxidized form of cysteine. Higher plasma levels of cystine are associated with increased risk of CVD
. Change in CD34+ Cell Count | Baseline, Month 6
  Cells expressing CD34 antigen (a protein encoded by the CD34 gene) are called CD34+ cells and can be isolated from blood samples. CD34+ cell count is a biomarker of regenerative capacity and reduced counts of CD34+ is associated with increased cardiovascular risk.
Change in Pulse Wave Velocity (PWV) | Baseline, Month 6
  Carotid-femoral artery pulse wave velocity (PWV) will be determined using transcutaneous Doppler flow velocity recordings simultaneously over the common carotid artery and the femoral artery. Aortic pulse wave velocity (PWV) estimates of the speed of the pressure wave traveling along the aorta and is regarded as a direct measure of large artery stiffness. Normal ranges for PWV are age based (PWV increases with age) and standardized thresholds for CVD risk have not been established. This study will assess the change in PWV in participants between baseline and after the 6 month intervention
Change in Reactive Hyperemia Index (RHI) | Baseline, Month 6
  Reactive Hyperemia Index (RHI) is a measure of microvascular endothelial function that is calculated as a ratio of preocclusion to postocclusion pulse signal amplitude. RHI will be estimated using digital pulse amplitude tonometry (EndoPAT). Greater RHI indicates better endothelial function.
Change in Glutathione | Baseline, Month 6
  Glutathione is a major antioxidant that helps eliminate peroxides and maintain cellular redox. Lower levels of glutathione are associated with cardiovascular disease.
Change in circulating progenitor cells (CPC) CD34+/CD133+ | Baseline, Month 6
  Progenitor cells (PCs), including CD34+/CD133+ cells, are part of the mechanisms underlying regeneration, and the pivotal role they play in vascular repair has only recently been appreciated. Endogenous PCs contribute to reendothelialization of tissues after endothelial injury, attenuating progression to frank atherosclerosis. Endothelial dysfunction correlates with PC number and function and a low PC count appears to be an independent predictor of poor outcome in patients with CAD, stroke or acute lung injury. CD34+/CD133+ cell counts improved risk prediction metrics beyond standard risk factors.
Change in circulating progenitor cells (CPCs) CD34+/VEGF2R+ | Baseline, Month 6
  Progenitor cells (PCs), including CD34+/VEGF2R+ cells, are part of the mechanisms underlying regeneration, and the pivotal role they play in vascular repair has only recently been appreciated. Endogenous PCs contribute to reendothelialization of tissues after endothelial injury, attenuating progression to frank atherosclerosis. Endothelial dysfunction correlates with PC number and function and a low PC count appears to be an independent predictor of poor outcome in patients with CAD, stroke or acute lung injury.
Change in Augmentation Index | Baseline, Month 6
  Augmentation index (AIx) is a composite measure of the magnitude of arterial wave reflections and systemic arterial stiffness and increases as the aortic pulse wave velocity (PWV) increases. Impaired arterial elastic properties, measured as the aortic AIx and/or PWV, are increasingly recognized as independent predictors of incident CVD events (myocardial infarction, stroke, revascularization), as well as all-cause mortality.
Change in Carotid Intima Media Thickness (CIMT) | Baseline, Month 6
  A CIMT scan is performed by using ultrasound determine the presence and severity of vascular disease. Presence of carotid plaque is associated with a 2-3-fold increased risk of future CVD events, and increased CIMT is associated with prevalent cardiovascular disease and an increased risk of myocardial infarction and stroke. Progression of CIMT has been used as a surrogate marker of change in CVD risk.

CONTACTS AND LOCATIONS:
Overall Officials: Herman Taylor, MD, Study Chair — Morehouse School of Medicine
Locations (2):
- United States (2):
  - Morehouse School of Medicine, Atlanta, Georgia
  - Emory University Clinical Research Network, Atlanta, Georgia

IPD SHARING:
Plan to Share IPD: No